CLINICAL TRIAL: NCT06801964
Title: Nutritional Supplementation in Patient With Stable COPD and in Those Recovering From an Acute Exacerbation of COPD: the Effects on Metabolism and Clinical Status
Brief Title: AECOPD and Nutritional Supplementation in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Associate Professor, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2014-0139
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Obstructive Pulmonary Disease; Exacerbation Copd
MeSH Terms: conditions — Lung Diseases, Obstructive | interventions — Proteins; Fish Oils; Olive Oil; Carbohydrates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AECOPD - No Nutrition (Experimental)
  Interventions: Other: Stable isotope infusion
- AECOPD - Nutrition (Experimental)
  Interventions: Other: Stable isotope infusion; Dietary Supplement: Protein and Fish Oil; Dietary Supplement: Protein and Olive Oil; Dietary Supplement: Carbohydrate and Olive Oil
- stable COPD (Experimental)
  Interventions: Other: Stable isotope infusion; Dietary Supplement: Protein and Fish Oil; Dietary Supplement: Protein and Olive Oil; Dietary Supplement: Carbohydrate and Olive Oil
- Healthy (Other)
  Interventions: Other: Stable isotope infusion

INTERVENTIONS:
Other: Stable isotope infusion — such as glycerol, D2O, tyrosine, phenylalanine, glucose, arginine, and citrulline
Dietary Supplement: Protein and Fish Oil — milk/carbohydrate mixture and supplementation of 3.5g of EPA+DHA (7g of fish oil)
  Arms: AECOPD - Nutrition; stable COPD
Dietary Supplement: Protein and Olive Oil — milk/carbohydrate mixture with olive oil
  Arms: AECOPD - Nutrition; stable COPD
Dietary Supplement: Carbohydrate and Olive Oil — carbohydrate mixture with olive oil
  Arms: AECOPD - Nutrition; stable COPD

SUMMARY:
Better understanding of the duration needed to overcome metabolic disturbances in patients experiencing exacerbation. Also, the explore role of nutritional intervention in the treatment program of stable COPD patients and in those recovering from an acute exacerbation (AECOPD) is important to restore loss of muscle mass and function and to reduce readmission and hospitalization rate of these patients, thereby leading to improved clinical and overall outcome as well as reduction of health care costs.

DETAILED DESCRIPTION:
Based on the literature, the Investigators hypothesize that an AECOPD is associated with an acute inflammatory response, accelerated muscle protein loss and compromised NO production and glutathione synthesis as compared to a stable COPD and healthy control group. Two weeks after AECOPD these disturbances are only partially restored and therefore nutritional intervention is required. Supplementation with milk proteins (containing essential amino acids) / carbohydrate (CHO) mixture in combination with fish oil supplementation will reduce the metabolic alterations in COPD patients recovering from an acute exacerbation but also in stable COPD as chronic systemic inflammation is also present in these patients. By simultaneously attenuating the catabolic effects of inflammation by fish oil and increasing the anabolic stimulus by high quality protein intake, muscle mass and function, will be restored, leading to better physical performance, condition and quality of life in COPD.

Specific aims:

* Specific aim 1: To test the hypothesis that AECOPD in outpatients results in severe net protein catabolism, impaired NO synthesis and GSH synthesis as compared to stable COPD. These disturbances are associated with impaired nutritional and functional status, and quality of life in COPD.
* Specific aim 2: To test the hypothesis that 14 days after AECOPD these disturbances are partially restored but still not comparable to that in stable chronic COPD patients and healthy control subjects. One group of participants with AECOPD will also be tested 10 weeks after exacerbation to see if metabolic disturbances have been restored.
* Specific aim 3: To test the effects of 8 weeks of nutritional supplementation with high-quality milk proteins (containing essential amino acids)/ carbohydrate (CHO) mixture with or without fish oil supplementation on protein and amino acid metabolism, muscle mass, muscle and cognitive function, physical performance, quality of life, and clinical and overall outcome in stable COPD patients and in those recovering from AECOPD.

ELIGIBILITY:
Inclusion criteria COPD exacerbation (AECOPD) group:

* Between age 45 and older
* Experiencing an acute exacerbation of COPD (defined as a combination of symptoms such as increased cough, sputum purulence, shortness of breath, systemic symptoms such as fever, and a decrease in FEV1 > 10% compared with values when clinically stable in the preceding years) and admitted at College Station Medical Center (with expected stay less than 10 days) or staying at home.
* Willingness and ability to comply with the protocol, including:
* Adhering to fasting state from 10 pm ± 2h onwards the day prior to each study visit
* Ability to lie in supine or elevated position for 4 hours

Inclusion criteria stable COPD subjects:

* Ability to walk, sit down and stand up independently
* Between age 45 and older
* Diagnosis of moderate to very severe chronic airflow limitation and compliant to the following criteria: FEV1 < 70% of reference FEV1
* Clinically stable condition and not suffering from a respiratory tract infection or exacerbation of their disease at least 4 weeks prior to the first test day
* Shortness of breath on exertion
* Willingness and ability to comply with the protocol, including:
* Adhering to fasting state from 10 pm ± 2h onwards the day prior to each study visit
* Ability to lie in supine or elevated position for 4 hours

Inclusion criteria healthy control subjects:

* Healthy male or female according to the investigator's or appointed staff's judgment
* Ability to walk, sit down and stand up independently
* Between age 45 and older
* No diagnosis of chronic airflow limitation
* Willingness and ability to comply with the protocol, including:
* Adhering to fasting state from 10 pm ± 2h onwards the day prior to each study visit
* Ability to lie in supine or elevated position for 4 hours

Exclusion Criteria all subjects:

* Any condition that may interfere with the definition 'healthy subject' according to the investigator's judgment (for healthy control group only)
* Established diagnosis of malignancy
* History of untreated metabolic diseases including hepatic or renal disorder
* Presence of other acute metabolic illnesses (ie renal, liver disease)
* Any other condition according to the PI or nurse that was found during the screening visit, that would interfere with the study or safety of the patient
* Dietary or lifestyle characteristics:
* Current alcohol or drug abuse
* Known hypersensitivity to fish and/or shellfish, Swanson EFAs Super EPA Fish oil or any of its ingredients, Swanson EFAs Certified Organic Extra Virgin Olive oil or any of its ingredients or Smartfish Nutrifriend or any of its ingredients (AECOPD and stable COPD nutrition groups only)
* Use of supplements containing more than 1 g of EPA+DHA 3 months prior to the first test day (AECOPD and stable COPD nutrition groups only)
* Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
* (Possible) pregnancy
* Body mass index <18.5 or >45 kg/m2
* When during the period from enrollment to completion of the study any condition is developed, whether causing a subject to not meet any of the inclusion criteria or to meet one or more of the exclusion criteria, the study can either be temporarily or permanently stopped for that subject.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Change in net whole-body protein synthesis | 2, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210 and 240 ± 5 minutes
  Change in whole-body protein synthesis rate

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Engelen, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No